CLINICAL TRIAL: NCT05058833
Title: Prospective Registry Evaluating Prognostic Impact of Cardiac Diastolic Function and Coronary Microvascular Function
Brief Title: Prognostic Impact of Cardiac Diastolic Function and Coronary Microvascular Function
Acronym: DIAST-CMD
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Collaborators: Chonnam National University Hospital (Other); Chosun University Hospital (Other); Gangneung Asan Hospital (Other)
Responsible Party: Principal Investigator, Joo Myung Lee, Assistant Professor, Samsung Medical Center
Other Study IDs: SMCDIAST119023
Record Dates: First submitted 2021-09-17; First posted 2021-09-28 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Ischemic Heart Disease; Microvascular Coronary Artery Disease; Diastolic Dysfunction; Heart Failure With Preserved Ejection Fraction
Keywords: coronary microvascular dysfunction; diastolic dysfunction; coronary flow reserve; index of microcirculatory resistance; prognosis
MeSH Terms: conditions — Myocardial Ischemia | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with cardiac diastolic dysfunction: Echocardiographic grades of diastolic function was defined according to 2016 ASE/EACVI recommendations for the evaluation of LV diastolic function. Cardiac diastolic dysfunction was defined as elevated E/e'≥15.
  Interventions: Diagnostic Test: Echocardiography; Diagnostic Test: Coronary flow reserve and index of microcirculatory dysfunction
- Patients with coronary microcirculatory dysfunction: Patients with coronary microcirculatory dysfunction was defined as having both depressed CFR (≤2.0) and elevated IMR (≥23U).
  Interventions: Diagnostic Test: Echocardiography; Diagnostic Test: Coronary flow reserve and index of microcirculatory dysfunction

INTERVENTIONS:
Diagnostic Test: Echocardiography — Echocardiographic grades of diastolic function was defined according to 2016 ASE/EACVI recommendations for the evaluation of LV diastolic function. Cardiac diastolic dysfunction was defined as elevated E/e'≥15.
Diagnostic Test: Coronary flow reserve and index of microcirculatory dysfunction — Coronary microcirculatory dysfunction was defined as having both depressed CFR (≤2.0) and elevated IMR (≥23U).

SUMMARY:
The DIAST-CMD registry (Prognostic Impact of Cardiac Diastolic Function and Coronary Microvascular Function) is prospective registry which enrolled patients who underwent echocardiography, cnically-indicated invasive coronary angiography and comprehensive physiologic assessments including fractional flow reserve (FFR), CFR, and IMR measurements for at least 1 vessel from Samsung Medical Center. Patients with hemodynamic instability, severe LV dysfunction (left ventricular ejection fraction<40%), a culprit vessel of acute coronary syndrome, severe valvular stenosis or regurgitation were excluded.

DETAILED DESCRIPTION:
Cardiac diastolic dysfunction refers to a condition in which abnormalities in mechanical function are present during diastole and is an independent predictor of mortality, even in patients with preserved left ventricular (LV) systolic function. Clinical manifestations of cardiac diastolic dysfunction are also variable, from asymptomatic subclinical heart failure to heart failure with preserved ejection fraction, angina or exercise intolerance without significant epicardial coronary artery disease, or end-stage heart failure. Although its pathophysiology remains incompletely understood, findings from clinical and pre-clinical studies have suggested systemic endothelial dysfunction, oxidative stress, and coronary microvascular dysfunction (CMD) could be important pathophysiologic mechanisms for cardiac diastolic dysfunction.

In this regard, recent studies evaluated non-invasively measured coronary flow reserve (CFR) from positron emission tomography (PET), cardiac magnetic resonance imaging (MRI), or Doppler echocardiography, and presented the association of depressed global CFR with cardiac diastolic dysfunction and higher risk of clinical events. The presence of CMD can be also evaluated by invasive physiologic assessment using both CFR and index of microcirculatory resistance (IMR). Previous studies presented CMD could be one of the major causes of angina without significant epicardial coronary artery disease and an independent predictor of adverse clinical events in patients with stable ischemic heart disease, acute myocardial infarction (MI), or myocardial disease. Nevertheless, there has been limited study which evaluated the association between cardiac diastolic dysfunction and CMD using invasive physiologic indices and their prognostic implications, especially in non-MI patients without significant coronary artery stenosis.

Therefore, the current study was designed the current DIAST-CMD registry to evaluate 3 important clinical questions as to whether: (1) cardiac diastolic dysfunction is significantly associated with the presence of CMD; 2) both cardiac diastolic dysfunction and CMD are significantly associated with long-term cardiovascular death; and 3) integration of both disease entities would have incremental prognostic stratification in non-MI patients without significant epicardial coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent clinically-indicated invasive coronary angiography
* Patients who underwent comprehensive physiologic assessments
* Patients who were evaluated by echocardiography

Exclusion Criteria:

* Patients with unavailable echocardiography data
* Patients with hemodynamic instability
* Patients with severe LV dysfunction (LV ejection fraction<30%)
* Patients with severe valvular stenosis or regurgitation
* Culprit vessel of acute coronary syndrome

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The DIAST-CMD registry (Prognostic Impact of Cardiac Diastolic Function and Coronary Microvascular Function) is prospective registry which enrolled patients who underwent echocardiography, cnically-indicated invasive coronary angiography and comprehensive physiologic assessments including fractional flow reserve (FFR), CFR, and IMR measurements for at least 1 vessel from Samsung Medical Center. Patients with hemodynamic instability, severe LV dysfunction (left ventricular ejection fraction<40%), a culprit vessel of acute coronary syndrome, severe valvular stenosis or regurgitation were excluded.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2016-04-08 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Cardiovascular death | 3 year
  Cardiovascular death

SECONDARY OUTCOMES:
all-cause death | 3 year
  all-cause death
Myocardial infarction | 3 year
  Myocardial infarction according to universal definition of MI
Any revascularization | 3 year
  Any revascularization according to ARC definition
Major adverse cardiac events | 3 year
  Major adverse cardiac events (MACEs, a composite of cardiovascular death, MI, and any revascularization)
Heart failure admission | 3 year
  Admission due to heart failure

CONTACTS AND LOCATIONS:
Overall Officials: Joo Myung Lee, MD, MPH, PhD, Principal Investigator — Samsung Medical Center
Locations (4):
- University of Iowa Carver College of Medicine, Iowa City, IA, USA, Iowa City, Iowa, United States
- South Korea (3):
  - Chonnam National University Hospital, Gwangju
  - Chosun University Hospital, Gwangju
  - Samsung Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: Undecided
The decision of sharing IPD will be determined after discussion by executive committee of the current study.

REFERENCES:
- [Derived] Lee SH, Choi KH, Hong D, Shin D, Joh HS, Kim HK, Park TK, Yang JH, Song YB, Hahn JY, Choi SH, Gwon HC, Lee JM. Prognostic Implications of Microvascular Resistance Reserve in Symptomatic Patients With Intermediate Coronary Stenosis. JACC Cardiovasc Interv. 2024 Mar 25;17(6):786-797. doi: 10.1016/j.jcin.2024.01.008. PMID 38538174
- [Derived] Hong D, Shin D, Lee SH, Joh HS, Choi KH, Kim HK, Ha SJ, Park TK, Yang JH, Song YB, Hahn JY, Choi SH, Gwon HC, Lee JM. Prognostic Impact of Coronary Microvascular Dysfunction According to Different Patterns by Invasive Physiologic Indexes in Symptomatic Patients With Intermediate Coronary Stenosis. Circ Cardiovasc Interv. 2023 Mar;16(3):e012621. doi: 10.1161/CIRCINTERVENTIONS.122.012621. Epub 2023 Feb 27. PMID 36846961
- [Derived] Hong D, Lee SH, Shin D, Choi KH, Kim HK, Ha SJ, Joh HS, Park TK, Yang JH, Song YB, Hahn JY, Choi SH, Gwon HC, Lee JM. Prognostic Impact of Cardiac Diastolic Function and Coronary Microvascular Function on Cardiovascular Death. J Am Heart Assoc. 2023 Feb 7;12(3):e027690. doi: 10.1161/JAHA.122.027690. Epub 2023 Jan 25. PMID 36695307
- [Derived] Chung YJ, Choi KH, Lee SH, Shin D, Hong D, Park S, Joh HS, Kim HK, Ha SJ, Park TK, Yang JH, Song YB, Hahn JY, Choi SH, Gwon HC, Lee JM. Prognostic Impact of Indeterminate Diastolic Function in Patients With Functionally Insignificant Coronary Stenosis. J Am Soc Echocardiogr. 2023 Mar;36(3):295-306.e5. doi: 10.1016/j.echo.2022.11.014. Epub 2022 Dec 5. PMID 36470507